CLINICAL TRIAL: NCT06015022
Title: Phase II Randomized Controlled Trial of Epigallocatechin Gallate for Hepatocellular Carcinoma Chemoprevention
Brief Title: EGCG for Hepatocellular Carcinoma Chemoprevention
Acronym: CATCH-B
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Yujin Hoshida, MD, PhD, Professor, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: STU-2023-0233
Record Dates: First submitted 2023-08-09; First posted 2023-08-29 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Cirrhosis, Liver
Keywords: hepatocellular carcinoma; chemoprevention; liver cancer
MeSH Terms: conditions — Liver Cirrhosis; Carcinoma, Hepatocellular; Liver Neoplasms | interventions — epigallocatechin gallate

STUDY DESIGN:
Intervention Model Description: Randomized placebo-controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Epigallocatechin gallate 600 - 800mg (Experimental): Epigallocatechin gallate (EGCG) 600mg will be administered daily via oral route for the initial 12 consecutive weeks on an outpatient basis. The dose of 600 mg will be continued for the second 12 weeks if an interim HCC biomarker test at the end of week 8 improves. If the interim test does not improve without dose-limiting adverse events, the dose will be increased to 800mg for the second 12 weeks, All participants will receive 24 weeks of treatment in total.
  Interventions: Drug: Epigallocatechin gallate (EGCG)
- Placebo (Placebo Comparator): Oral administration of placebo for 24 weeks
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Epigallocatechin gallate (EGCG) — EGCG is a green tea-derived catechin
  Other Names: Teavigo
  Arms: Epigallocatechin gallate 600 - 800mg
Other: Placebo — Placebo in the same capsule with the experimental agent (EGCG).
  Arms: Placebo

SUMMARY:
This phase II trial tests epigallocatechin gallate (EGCG) for its efficacy and safety in preventing development of hepatocellular carcinoma (HCC) in patients with liver cirrhosis.

DETAILED DESCRIPTION:
This study will evaluate whether EGCG favorably modulate an HCC risk biomarker (PLSec) with acceptable safety profile in patients with compensated cirrhosis and elevated HCC risk determined by clinical variable-based score (FIB-4 index) and PLSec. Sixty participants will be randomized (1:1) to either the study drub or placebo arm and receive the treatment for 24 weeks. The participants will orally take EGCG 600 mg capsules or placebo for the first 12 weeks. If an interim PLSec analysis at the end of week 8 is not improved without any dose-limiting adverse events, the dose will be increased to 800 mg for the second 12 weeks. If the interim PLSec is improved, 600 mg will be continued. After completing the 24-week treatment, change in the PLSec test with the treatment is calculated by comparing pre- and post-treatment serum samples in each patient, and the changes will be compared between the treatment arms (primary endpoint). Complete adverse event profiles will be recorded, and change in quality of life will be compared between the treatment arms (secondary endpoints). If optional paired liver biopsy tissues are obtained, changes in tissue-based HCC risk biomarker (PLS) and immunohistochemical markers of cell proliferation, neoplasm, senescence, and fibrogenesis will be determined, changes in the FIB-4 index and liver stiffness measurement will be determined, and association with incident HCC during the study period will be evaluated (exploratory endpoints).

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥ 18 years-old)
* Clinically and/or histologically diagnosed cirrhosis
* No active hepatic decompensation
* No prior history of HCC
* Adequate hematologic, hepatic, and renal function
* Karnofsky performance status score ≥70
* Both sexes and all racial/ethnic groups will be considered
* FIB-4 index > 3.25
* High-risk PLSec at baseline
* Absence of HLA-B*35:01

Exclusion Criteria:

* Prior or ongoing use of EGCG
* History of adverse reaction to green tea products
* Severe obesity (BMI > 40 kg/m2)
* Active drinking
* EGCG treatment <4 weeks or <80% of planned regimen at the end of week 4
* HCC development during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2028-08-31 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
Change in Prognostic Liver Secretome signature (PLSec) score | Baseline to week 24
  HCC risk level at baseline and post-treatment will be determined as Prognostic Liver Secretome signature (PLSec) score, ranging from 0 (lowest risk) to 8 (highest risk).
  Change in the biomarker-based HCC risk level will be calculated as delta-PLSec by subtracting the post-treatment PLSec score from the baseline pre-treatment PLSec score. delta-PLSec values will be compared between the EGCG and placebo arms using two-sample t-test.

SECONDARY OUTCOMES:
Complete adverse event profile | Baseline to week 24
  Adverse events are monitored at least monthly and graded/recorded according to National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) version 5. The number and severity of adverse events will be tabulated and summarized across all grades. Grade 3+ adverse events will be similarly described and summarized separately.
Change in quality of life measured by the chronic liver disease questionnaire | Baseline to week 24
  Quality of life (QOL) will be measured by using the chronic liver disease questionnaire (CLDQ), which consists of 29 questions. Participants can select one answer from seven choices of descriptive answers for each question. Frequency distributions, graphical techniques and other descriptive measures will be used to summarize the results. When frequencies are compared, Fisher's exact test will be used.

OTHER OUTCOMES:
Change in hepatic gene expression-based HCC risk biomarker, Prognostic Liver Signature (PLS) (optional) | Baseline to week 24
  When optional liver biopsy tissue is obtained, modulation of hepatic gene expression-based signature associated with HCC risk, Prognostic Liver Signature (PLS) is measured by comparing pre- and post-treatment liver biopsy samples. Change in HCC risk level will be quantified as combined enrichment score (CES) by comparing between the 2 time points. A positive and negative CES values indicate worsening and improvement of the PLS, respectively. Absolute value of the CES indicate magnitude of reduction (i.e., negative value) or increase (i.e., positive value) of HCC risk level. There is no defined range of CES. CES values are compared between the EGCG and placebo arms using two-sample t-test.
Change in positive signal intensities of immunohistochemistry markers (optional) | Baseline to week 24
  When optional liver biopsy tissue is obtained, change of immunohistochemical markers of cellular proliferation (Ki67), hepatic neoplasia (GST-p), cellular senescence (beta-gal), fibrogenesis (alpha-SMA) will be assessed using formalin-fixed pre-treatment paraffin-embedded (FFPE) tissues. Positivity for all of the markers will be quantified by higher intensity at pixel levels in captured images using the ImageJ software. The measurements are compared between the EGCG and placebo arms using one-sample t-test.
HCC incidence | Average time frame of 1 year
  The participants will be regularly followed every 6 months for HCC development for their life time. HCC diagnosis is based on the American Association for Study of Liver Disease (AASLD) clinical practice guidelines. Time to HCC development will be calculated as days between the treatment initiation data and date of HCC diagnosis. Cumulative HCC incidence will be compared between the treatment arms using log-rank test and Cox regression within and beyond the study period. This exploratory analysis will be performed through study completion with an anticipated average time frame of 1 year.

CONTACTS AND LOCATIONS:
Overall Officials: Yujin Hoshida, MD, PhD, Principal Investigator — UT Southwestern
Locations (1):
- UT Southwestern, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No